CLINICAL TRIAL: NCT00628706
Title: Investigating the Acute Effects of THC on Functional Brain Systems
Acronym: FIX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Center for Human Drug Research (Unknown); Leiden University Medical Center (Other); TI Pharma (Unknown)
Responsible Party: Prof. N.F. Ramsey, UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: THC-phMRI-01
Record Dates: First submitted 2008-02-24; First posted 2008-03-05 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Reward; Tetrahydrocannabinol; Endocannabinoids; Memory; Magnetic Resonance Imaging
Keywords: tetrahydrocannabinol; memory; reward; magnetic resonance imaging; endocannabinoids
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Inhalation of THC, using a Volcano vaporizer
  Interventions: Drug: Delta9-tetrahydrocannabinol (THC)
- B (Placebo Comparator): Inhalation of vehicle, using a Volcano vaporizer
  Interventions: Drug: Delta9-tetrahydrocannabinol (THC)

INTERVENTIONS:
Drug: Delta9-tetrahydrocannabinol (THC) — inhalation of 6 mg liquid THC, vaporized by means of a Volcano vaporizer
  Other Names: dronabinol, marinol, THC, tetrahydrocannabinol

SUMMARY:
The purpose of this study is to determine whether THC, the main psychoactive ingredient in cannabis, affects functional brain systems underlying memory and reward.

DETAILED DESCRIPTION:
Cannabis is by far the most frequently used illicit drug worldwide and has significant effects on memory. Further, cannabis has an addictive potential. These effects are mediated by an action of THC, the main psychoactive ingredient of cannabis, on cannabinoid CB1 receptors. These receptors are particularly highly expressed in brain regions involved in memory and reward. Therefore, in this study we will investigate the acute effects of THC on functional brain systems underlying memory and reward. We will visualize these effects using the latest non-invasive imaging technique: pharmacological MRI (phMRI).

ELIGIBILITY:
Inclusion Criteria:

* History of mild cannabis use for at least one year (<1/week and ≥ 4/year)
* History without psychotic experiences after cannabis use
* Age between 18 and 45 years
* Right-handedness, assessed with the Edinburgh Handedness Inventory
* Written informed consent of the subject

Exclusion Criteria:

* Any clinical significant abnormality of any clinical laboratory test, including urinary drug screening
* Impaired physical health evaluated by medical history, physical (including neurological) examination and screening laboratory tests
* History of clinically significant psychiatric or neurological illness
* History of clinically significant psychiatric or neurological illness in first- or second-degree relatives
* History of alcohol and/or drug abuse (DSM-IV criteria)
* Body Mass Index (B.M.I.) <18 kg/m2 or >28 kg/m2
* Paranoid ideation or psychoticism on SCL-90
* Any subject who received any investigational medication within 90 days prior to the start of the study or who is scheduled to receive an investigational drug
* The use of any medication within three weeks prior to the start of the study, except for paracetamol
* Positive HIV or Hepatitis B/C test
* Blood donation within 3 months before the start of the study
* Claustrophobia
* Metal objects in or around the body (braces, pacemaker, metal fragments)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The main study parameter is the blood oxygen level dependent (BOLD) signal. | 4 months

SECONDARY OUTCOMES:
Behavioral parameters (two VAS questionnaires) | 4 months
Cerebral blood flow (ASL) | 4 months
Concentration of plasma THC and its main metabolites | 4 months
Performance on neuropsychological tests | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Nick Ramsey, Professor, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Bossong MG, Jager G, van Hell HH, Zuurman L, Jansma JM, Mehta MA, van Gerven JM, Kahn RS, Ramsey NF. Effects of Delta9-tetrahydrocannabinol administration on human encoding and recall memory function: a pharmacological FMRI study. J Cogn Neurosci. 2012 Mar;24(3):588-99. doi: 10.1162/jocn_a_00156. Epub 2011 Nov 8. PMID 22066583